CLINICAL TRIAL: NCT03703765
Title: Volume Estimation of Lower Limbs Before and After Endovascular Venous Intervention or Conventional Surgery in Venous Disease
Brief Title: Volume Estimation of the Limb After VEnous Treatment
Acronym: VELVET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-A02698-45
Record Dates: First submitted 2018-01-18; First posted 2018-10-12 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Venous Disease
Keywords: Volume; veins; lower limb; imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lower limb volume estimation (Experimental): Patients referred for a preoperative venous assessment as part of an indication for interventional management, whether by conventional or endovascular surgery, of a chronic venous pathology.
  Intervention is measurement of lower limb volume with scanner 3D system before and after surgery or vascular intervention.
  Interventions: Device: lower limb volume estimation

INTERVENTIONS:
Device: lower limb volume estimation — The 3D scanner system is a three-dimensional measurement system.
  It allows to evaluate the volume of the lower limbs in order to quantify the evolution of the edema of the lower limbs in the venous pathology in pre and post therapeutic technique.
  It is a non-invasive, easily accepted, non-invasive, non-invasive technique that minimizes discomfort.

SUMMARY:
Chronic venous disease encompasses a broad spectrum of clinical presentations and is considered the most common vascular disease. Its causes are diverse, including primary defects of the wall or valves, chronic venous insufficiency, or lesions secondary to thrombosis, a post-thrombotic venous disease, affecting the superficial or deep venous network or both. The major symptom of venous disease is the enlargement of the lower limbs, which can result in edema. The evaluation of the volume of the lower limbs is very important in the diagnosis and follow-up of the venous pathology. There is a great variability of clinical pictures making it difficult to choose the therapeutic gesture. Endovascular venous interventions and conventional venous surgery are major advances in the treatment of venous disease. The variation of lower limb volume in pre and post procedure is a determining factor; thus orienting clinicians for post interventional therapeutic monitoring. Indeed the management of venous disease is multidisciplinary, it involves the cooperation of several specialists as part of its monitoring and its therapeutic management. Our collaborative group includes the Adult and Child Vascular Investigations Department, the Vascular Clinic, the Cardiovascular and Thoracic Surgery Department, and the Interventional Radiology Department. The evaluation of the variation of the volumes of the lower limbs is a capital data for the various specialists for the care in pre and post procedure. A volumetric 3D scanner system guarantees a reliable measurement ensuring optimal evolution and therapeutic follow-up.

DETAILED DESCRIPTION:
At admission eligible patients are proposed to participate. Written consent is signed after complete oral and written explanation of the protocol is signed. No register of non-included patients will be kept.

In included patients, in parallel to the routine ultrasound investigation for which the patient is referred, the evaluation of the variation of the volumes of the lower limbs with the volumetric 3D scanner will be performed as explained later in arm description.

Usual ongoing treatments are obtained by history and recorded. The end of the visit is the end of the participation of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* subjects referred for investigation of a preoperative venous assessment
* affiliation to the French National healthcare system
* french speaking patients

Exclusion Criteria:

* pregnancy
* inability to understand the study goal
* patients protected by decision of law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Volume of lower limbs | 12 months
  Change of volume of the lower limbs will be assessed with a volumetric 3D scanner

SECONDARY OUTCOMES:
Change in symptoms and quality of life | 12 months
  Change in symptoms and quality of life of patients assessed with the CIVIQ questionnaire
Change in symptoms and quality of life | 12 months
  Change in symptoms and quality of life of patients assessed with the SF36 questionnaire
Change in symptoms and quality of life | 12 months
  Change in symptoms and quality of life of patients assessed with the Villalta score for patients treated for post thrombotic syndrome
Change in symptoms and quality of life | 12 months
  Change in symptoms and quality of life of patients assessed with the CEAP classification for patients treated for superficial venous insufficiency
Validity | 1 hour
  To validate the measurement of the volume of the lower limbs by a 3D scanner system compared to measurement by a tape measure (gold standard) in venous disease.

CONTACTS AND LOCATIONS:
Overall Officials: HENNI MD SAMIR, PhD, Principal Investigator — University Hospital, Angers
Locations (1):
- UH Angers, Angers, France

IPD SHARING:
Plan to Share IPD: Undecided